CLINICAL TRIAL: NCT01409941
Title: The Prognostic Relevance of N-terminal Pro B-type Natriuretic Peptide(NTproBNP), Cerebral Oxygen Saturation (ScO2), and Preoperative Creatinine Clearance in Cardiac Surgery Patients - Amendment 2: the Role of NTproBNP and ScO2 in Predicting Mortality and Postoperative Organ Dysfunction.
Brief Title: The Relation Between Preoperative ScO2 and the Postoperative Course of Humoral Organ Dysfunction Markers.
Status: Completed | Type: Observational
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Matthias Heringlake, Prof. Dr. med. Matthias Heringlake, University of Luebeck
Other Study IDs: CS_RS_2008-2009 - ScO2
Record Dates: First submitted 2011-08-03; First posted 2011-08-04 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Patients Undergoing Cardiac Surgery
Keywords: cerebral oxygen saturation,; NTproBNP; hsTNT; GDF-15

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and urinary samples.
Oversight: Data Monitoring Committee: No

SUMMARY:
Cerebral oxygen saturation (ScO2) is a measure of cerebral and systemic oxygen delivery to demand ratio. An observational trial in a heterogeneous cohort of 1078 patients patients revealed that a ScO2 below 50% absolute during oxygen insufflation is an independent predictor of short and long term mortality in patients undergoing on-pump cardiac surgery. Comparably, a low ScO2 was a predictor of postoperative morbidity determined as a combined endpoint of a high dependency unit stay of more than 9 days and/or at least 2 of the major postoperative complications. low cardiac output syndrome, stroke, need of renal replacement therapy or reintubation.

The primary objectives of the present prospective observational study is to determine, if there is an association between preoperative ScO2 and postoperative organ dysfunction determined by sensitive markers of organ dysfunction (N-Terminal pro B-type natriuretic peptide, high sensitive troponin T, growth-differentiation factor 15, soluble -FLT1, and placental growth factor)

ELIGIBILITY:
Inclusion Criteria:

* all patients scheduled for cardiac surgery

Exclusion Criteria:

* age less than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for cardiac surgery
Sampling Method: Probability Sample
Enrollment: 765 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Mortality | 1 year

SECONDARY OUTCOMES:
Morbidity | Within hospital

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Heringlake, MD, Principal Investigator — Department of Anesthesiology, University of Luebeck